CLINICAL TRIAL: NCT06968221
Title: A Study on the Safety and Efficacy of Using Cingular Bovine Pericardium Anastomosis Reinforcement Membrane for Tissue Reinforcement and Hemostasis at Anastomotic Sites
Brief Title: Bovine Reinforcement in Stomach, Colorectal and Lung Operation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Cingularbio Co. Ltd (Industry)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSLR-2024-01
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer Stage III; Lung Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: with a bioabsorbable staple line reinforcement material compared with standard non-reinforced material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioabsorbable Staple Line Reinforcement configured for circular staplers (Experimental): stomach, Colorectal and lung anastomotic staple line reinforcement with Bioabsorbable Staple Line Reinforcement configured for circular staple
  Interventions: Device: Bioabsorbable Staple Line Reinforcemen
- anastomotic staple line without reinforcement (Active Comparator): stomach, colorectal and lung anastomotic staple line without reinforcement
  Interventions: Device: Bioabsorbable Staple Line Reinforcemen

INTERVENTIONS:
Device: Bioabsorbable Staple Line Reinforcemen — cingular Bioabsorbable Staple Line Reinforcement

SUMMARY:
The primary purpose of this prospective, randomized multicenter center study is to evaluate and compare the outcomes of stomach,colorectal and lung anastomoses reinforced with a bioabsorbable staple line reinforcement material compared with standard non-reinforced techniques with respect to the incidence of postoperative hemorrage rate, anastomotic leakage, if applicable.

DETAILED DESCRIPTION:
This is a randomized prospective trial that compares the use of Cingular Bioabsorbable Staple Line Reinforcement to standard stapling techniques in tissue resections. The potential exists to utilize staple line reinforcement as a means of lowering the rate of post-operative hemorrage rate, anastomotic leakage.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will undergo operation with stapled stomach, colorectal anastomosis with or without reinforcement
* Subjects willing to accept informed consent and willing to attend the follow up

Exclusion Criteria:

* Subjects who have significant intraoperative hypotension or cardiac events.
* Subjects with collagen vascular disease, coagulopathy, significant renal or hepatic dysfunction (creatinine >1.6 or liver enzymes > 50% upper limit of normal values).
* Subjects have uncontrolled intra-abdominal infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects Who Experience a hemorrage | 10 min
  The primary endpoint for the study is the proportion of subjects who experience a hemorrage through 10 min post procedure.

SECONDARY OUTCOMES:
Proportion of Subjects Who Experience a Clinical and/or Radiologic Anastomotic Leak | 1-3 months
  The primary endpoint for the study is the proportion of subjects who experience a clinical and/or radiologic anastomotic leak through 1-3 months post procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hospital affiliated to Shanghai jiaotong Uni school of medicine, Shanghai, China